CLINICAL TRIAL: NCT04271592
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single and Multiple Dose Escalation and Food Effect Study of ABI-H3733 in Healthy Subjects
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of ABI-H3733 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-H3733-101; U1111-1246-2965 (Other: World Health Organization)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part 1: SAD Cohorts 1-7 ABI-H3733 Liquid Form (Experimental): A single dose of ABI-H3733 liquid oral dosage form administered on Day 1. Cohort 1 will receive a 100-mg dose. Subsequent cohorts 2-7 will receive a ≤3-fold increase in dose from the previous cohort; the dose will be determined by evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: ABI-H3733 Liquid Oral Dosage Form
- Part 1: SAD Cohorts 1-7 Placebo Liquid Form (Placebo Comparator): A single dose of placebo matching ABI-H3733 liquid oral dosage form will be administered on Day 1. Cohort 1 will receive a 100-mg dose. Subsequent cohorts 2-7 will receive a ≤3-fold increase in dose from the previous cohort; the dose will be determined by evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: Placebo to ABI-H3733 Liquid Oral Dosage Form
- Part 1: MAD Cohorts 8-10 ABI-H3733 Liquid Form (Experimental): Once-daily doses of ABI-H3733 liquid oral dosage form will be administered from Day 1 to Day 5. Cohort 8 will receive a dose determined from evaluation of the data from the SAD cohorts. Subsequent cohorts 9 and 10 will receive a ≤3-fold increase in dose from the previous cohort; the dose will be determined by evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: ABI-H3733 Liquid Oral Dosage Form
- Part 1: MAD Cohorts 8-10 Placebo Liquid Form (Placebo Comparator): Once-daily doses of placebo matching ABI-H3733 liquid oral dosage form will be administered from Day 1 to Day 5. Cohort 8 will receive a dose determined from evaluation of the data from the SAD cohorts. Subsequent cohorts 9 and 10 will receive a ≤3-fold increase in dose from the previous cohort; the dose will be determined by evaluation of safety and PK data from previous cohorts.
  Interventions: Drug: Placebo to ABI-H3733 Liquid Oral Dosage Form
- Part 2: Single Dose Fasted Cohort 11 ABI-H3733 Solid Form (Experimental): A single dose of ABI-H3733 solid oral dosage form will be administered in a fasted state on Day 1. The decision to proceed with Part 2 and the dose administered will be determined after evaluation of cumulative safety and PK data from Part 1.
  Interventions: Drug: ABI-H3733 Solid Oral Dosage Form
- Part 2: Single Dose Fasted Cohort 11 Placebo Solid Form (Placebo Comparator): A single dose of placebo matching ABI-H3733 liquid oral dosage form will be administered in a fasted state on Day 1. The decision to proceed with Part 2 and the dose administered will be determined after evaluation of cumulative safety and PK data from Part 1.
  Interventions: Drug: Placebo to ABI-H3733 Solid Oral Dosage Form
- Part 2: Single Dose Fed Cohort 12 ABI-H3733 Solid Form (Experimental): A single dose of ABI-H3733 solid oral dosage form will be administered after a high-fat meal on Day 1. The decision to proceed with Part 2 and the dose administered will be determined after evaluation of cumulative safety and PK data from Part 1.
  Interventions: Drug: ABI-H3733 Solid Oral Dosage Form
- Part 2: Single Dose Fed Cohort 12 Placebo Solid Form (Placebo Comparator): A single dose of placebo matching ABI-H3733 solid oral dosage form will be administered after a high-fat meal on Day 1. The decision to proceed with Part 2 and the dose administered will be determined after evaluation of cumulative safety and PK data from Part 1.
  Interventions: Drug: Placebo to ABI-H3733 Solid Oral Dosage Form

INTERVENTIONS:
Drug: ABI-H3733 Liquid Oral Dosage Form — ABI-H3733 liquid oral dosage form
  Arms: Part 1: MAD Cohorts 8-10 ABI-H3733 Liquid Form; Part 1: SAD Cohorts 1-7 ABI-H3733 Liquid Form
Drug: ABI-H3733 Solid Oral Dosage Form — ABI-H3733 solid oral dosage form
  Arms: Part 2: Single Dose Fasted Cohort 11 ABI-H3733 Solid Form; Part 2: Single Dose Fed Cohort 12 ABI-H3733 Solid Form
Drug: Placebo to ABI-H3733 Liquid Oral Dosage Form — Placebo to ABI-H3733 liquid oral dosage form
  Arms: Part 1: MAD Cohorts 8-10 Placebo Liquid Form; Part 1: SAD Cohorts 1-7 Placebo Liquid Form
Drug: Placebo to ABI-H3733 Solid Oral Dosage Form — Placebo to ABI-H3733 solid oral dosage form
  Arms: Part 2: Single Dose Fasted Cohort 11 Placebo Solid Form; Part 2: Single Dose Fed Cohort 12 Placebo Solid Form

SUMMARY:
This study is designed to assess safety, tolerability, pharmacokinetics (PK), formulation (liquid and solid oral forms) and food effect of ABI-H3733 in healthy participants. Part 1 includes evaluation of the safety, tolerability, and PK of ABI-H3733 during single ascending dose (SAD) and multiple-ascending dose (MAD) administration of the oral liquid formulation. Part 2 includes assessment of a solid dosage formulation of ABI-H3733 in participants under fasted conditions or after a high-fat meal. Optional cohorts may be enrolled in Parts 1 and 2 of the study to explore additional dose levels, solid oral dosage formulations, or for cohort expansion.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, medical history, or clinical laboratory results at screening.

Exclusion Criteria:

* Positive test results for human immunodeficiency virus (HIV) or hepatitis B or C.
* History of or current persistent drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events | Up to Day 10
Number of Participants with One or More Related Adverse Events | Up to Day 10
Number of Participants with One or More Severe (Grade ≥3) Adverse Events | Up to Day 10

SECONDARY OUTCOMES:
SAD Cohorts 1-7: Area Under the Plasma Concentration Time Curve (AUC) of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
SAD Cohorts 1-7: Maximum Plasma Concentration (Cmax) ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
SAD Cohorts 1-7: Time of Cmax (Tmax) of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
SAD Cohorts 1-7: Apparent Terminal Elimination Half-life (t1/2) of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
SAD Cohorts 1-7: Apparent Systemic Clearance (CL/F) of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
SAD Cohorts 1-7: Apparent Volume of Distribution (Vz/F) of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
MAD Cohorts 8-10: AUC of ABI-H3733 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before and up to 120 hours after dosing on Day 5
MAD Cohorts 8-10: Cmax Over the Dosing Interval of ABI-H3733 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before and up to 120 hours after dosing on Day 5
MAD Cohorts 8-10: Tmax of ABI-H3733 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before and up to 120 hours after dosing on Day 5
MAD Cohorts 8-10: t1/2 of ABI-H3733 | before and at pre-specified time points up to 24 hours after dosing on Day 1; before and up to 120 hours after dosing on Day 5
Single Dose Cohorts 11-12: AUC of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
Single Dose Cohorts 11-12: Cmax of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
Single Dose Cohorts 11-12: Tmax of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing
Single Dose Cohorts 11-12: t1/2 of ABI-H3733 | before and at pre-specified time points up to 120 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Katia Alves, MD, Study Director — Assembly Biosciences
Locations (1):
- Auckland Clinical Studies, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No